CLINICAL TRIAL: NCT07218120
Title: A Randomized Trial of Financial Incentives for In-Person Recruitment of Individuals to the Alzheimer's Prevention Trial (APT) Webstudy
Brief Title: In-Person Recruitment of Individuals to the Alzheimer's Prevention Trial (APT) Webstudy
Acronym: FIND-AD Aim 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Vision y Compromiso (Unknown); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Mireille Jacobson, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-24-01201; 964386, 946223 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-10-10; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-06

CONDITIONS: Memory Decline; Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial incentive (Experimental): Participants in this arm will receive a gift card for enrolling in the APT Web Study
  Interventions: Other: Financial Incentive
- Nominal value gift (Active Comparator): Participants in this arm will receive a $0-$2 gift for enrolling in the APT Web Study.
  Interventions: Other: Active Comparator #1

INTERVENTIONS:
Other: Financial Incentive — $25 gift card
  Arms: Financial incentive
Other: Active Comparator #1 — Nominal value gift
  Arms: Nominal value gift

SUMMARY:
Women, older adults, individuals from communities of color, particularly Black and Latino persons, and individuals with lower socioeconomic status are historically underrepresented in clinical research. This is true across a range of clinical areas but no more so than in Alzheimer's Disease Research. The purpose of this study is to assess whether offering small $25 financial incentives can increase enrollment of diverse community members to the Alzheimer's Prevention Trial (APT) Webstudy, a memory concerns registry meant to accelerate clinical trials, relative to non-monetary incentives such as a reusable grocery bag. To do this we will test in-person recruitment efforts at community events and locations, such as Northgate Gonzalez Market locations and local food bank events. We also aim to compare the relative cost of recruiting an additional person to the APT Webstudy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 and over.
* Able to read English or Spansih
* Email access

Exclusion Criteria:

* Current dementia diagnosis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
APT Webstudy Enrollment | Day 1
  Participant enrolled in the APT Webstudy, which includes completion of at least one of two remote cognitive assessments, on the recruitment day.

SECONDARY OUTCOMES:
Completion of both cognitive assessments | Day 1
  Completion of both APT Webstudy cognitive assessments - the CFI and the BRANCH.
Cost per enrollee | Day 1
  Cost per additional enrollee by arm

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Jaocbson, PhD, Principal Investigator — University of Southern California
Locations (1):
- Northgate Gonzalez Market, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Age, Language, Location, Date, Randomization Status, Enrollment Status
Supporting Information: Study Protocol